CLINICAL TRIAL: NCT06941909
Title: THE EFFECT OF A MINDFULNESS-BASED SELF-COMPASSION PROGRAM ON CARE BURDEN, LIFE SATISFACTION, AND COPING LEVELS OF CAREGIVERS OF INDIVIDUALS WITH SCHIZOPHRENIA: A RANDOMIZED CONTROLLED TRIAL PROTOCOL
Brief Title: The Effect of a Mindfulness-Based Self-Compassion Program on Care Burden, Life Satisfaction, and Coping Levels of Caregivers of Individuals With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neslihan Lok (Other)
Responsible Party: Sponsor-Investigator, Neslihan Lok, Prof. Dr., Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-BK-01; 23212021 (Other Grant/Funding Number: Selcuk University BAP project)
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Care Givers; Burden, Caregiver; Stress; Satisfaction With Life
Keywords: Care burden; Mindfulness-Based Self-Compassion Programme; Life Satisfaction; Coping with Stress; Schizophrenia.
MeSH Terms: conditions — Caregiver Burden; Personal Satisfaction; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants in the intervention group received weekly online group training and counseling sessions for a duration of 8 weeks. After each session, participants were provided with a practice guide and audio recordings to support home practice.
  Interventions: Other: Mindfulness-Based Self-Compassion
- control group (No Intervention): The control group did not receive any intervention during the study period.

INTERVENTIONS:
Other: Mindfulness-Based Self-Compassion — The intervention consisted of weekly online group training and counseling sessions over an 8-week period. Following each session, participants were provided with a practice guide and audio recordings to support home-based practice.
  Other Names: Mindfulness-Based Self-Compassion Program
  Arms: intervention group

SUMMARY:
This study aims to examine the effect of the Mindfulness-Based Self-Compassion Program on caregiver burden, life satisfaction, and coping with stress levels among caregivers of individuals diagnosed with schizophrenia. This is a randomized controlled trial with a parallel-group design. The study sample consists of caregivers of individuals diagnosed with schizophrenia who have applied to the psychiatry outpatient clinic of a university hospital within the past year. Caregivers who meet the inclusion criteria will be randomly assigned to intervention and control groups. The program was delivered over eight weeks through group training and counseling sessions. The findings of this study are expected to guide the development of interventions targeting caregiver burden, life satisfaction, and coping strategies among caregivers.

Research Hypotheses H1.1: The caregiver burden of the intervention group receiving the Mindfulness-Based Self-Compassion Program is lower than that of the control group.

H1.2: The life satisfaction of the intervention group receiving the Mindfulness-Based Self-Compassion Program is higher than that of the control group.

H1.3: The coping level of the intervention group receiving the Mindfulness-Based Self-Compassion Program is higher than that of the control group.

H1.3.1: The self-confident coping approach of the intervention group is higher than that of the control group.

H1.3.2: The optimistic coping approach of the intervention group is higher than that of the control group.

H1.3.3: The tendency to seek social support in the intervention group is higher than in the control group.

H1.3.4: The helpless coping approach of the intervention group is lower than that of the control group.

H1.3.5: The submissive coping approach of the intervention group is lower than that of the control group.

DETAILED DESCRIPTION:
In this randomized controlled trial, the effect of the Mindfulness-Based Self-Compassion Program on caregiver burden, life satisfaction, and coping styles of individuals providing care for people diagnosed with schizophrenia was evaluated. The study was designed with a parallel-group structure consisting of an intervention and a control group.

The sample size was calculated using the G*Power 3.1.9.4 software at a 95% confidence level. Based on the mean scores of the Functional Recovery Scale from a previous study, a total of 40 participants (20 in each group) were determined to be sufficient, with 80% power, an effect size of 0.9237531, and a 5% margin of error. To account for potential attrition, the sample size was increased by 10%, and the study was completed with 44 participants.

Caregivers who met the inclusion and exclusion criteria and voluntarily agreed to participate were randomly assigned to the intervention and control groups using a simple randomization method performed by an independent statistician. This approach was chosen to minimize selection bias and control for potential confounding variables.

Participants in the intervention group received weekly online group training and counseling sessions for a duration of 8 weeks. After each session, participants were provided with a practice guide and audio recordings to support home practice. The control group did not receive any intervention during the study period.

Pre-tests and informed consent were obtained prior to randomization, while post-tests were conducted by the researchers at the end of the 8-week program. Upon completion of data collection, the Mindfulness-Based Self-Compassion Program was also offered to the control group.

The program was based on the theoretical framework developed by Germer and Neff (2019) and Neff and Germer (2018), and structured as an eight-week curriculum centered around the concepts of mindfulness and self-compassion. Each session lasted approximately 90 minutes and was conducted once a week.

The content of the program was developed based on existing literature and training materials. Expert opinions were sought during the development process, including feedback from six faculty members-three from psychiatric nursing, two from public health nursing, and one from the field of guidance and psychological counseling. The final version of the program was shaped in accordance with these expert recommendations.

The primary outcome variables of the study were caregiver burden, life satisfaction, and coping styles. Data were collected using the Personal Information Form, Zarit Burden Interview, Satisfaction with Life Scale, and Coping Styles Inventory

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older and providing care for an individual diagnosed with schizophrenia according to ICD-10 criteria
* The care recipient must be registered with the Psychiatry Outpatient Clinic of Selçuk University Faculty of Medicine Hospital and attend regular follow-up appointments
* Providing care for a period of at least 3 months within the last year
* Having access to a mobile phone or computer to participate in online sessions

Exclusion Criteria:

* Having a diagnosed organic mental disorder
* Having any chronic psychiatric illness
* Experiencing hearing, comprehension, or speech impairments
* Concurrent participation in a similar intervention program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-01-13 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Change in caregiver burden (Zarit Caregiver Burden Scale) | Baseline and 8 weeks after the intervention
  Caregiver burden levels will be assessed using the Zarit Caregiver Burden Scale. Higher scores indicate greater burden. Comparison will be made between baseline and 8th week post-intervention.
Change in life satisfaction as measured by the Satisfaction with Life Scale (SWLS) | Baseline and 8 weeks post-intervention
  This outcome evaluates the effect of the Mindfulness-Based Self-Compassion Program on life satisfaction levels among caregivers of individuals diagnosed with schizophrenia. The SWLS will be used to assess participants' perceptions of life satisfaction at baseline and post-intervention.
Change in coping strategies as measured by the Coping Styles Inventory | Baseline and 8 weeks after the intervention
  This outcome examines changes in coping styles (self-confident, optimistic, seeking social support, helpless, and submissive) in caregivers who participate in the Mindfulness-Based Self-Compassion Program. The Coping Styles Inventory will be administered before and after the program to assess differences in adaptive and maladaptive coping strategies.

SECONDARY OUTCOMES:
Change in self-confident coping style | Baseline and 8 weeks after the intervention
  This secondary outcome evaluates the change in the use of self-confident coping strategies among caregivers following participation in the Mindfulness-Based Self-Compassion Program. Measured using the self-confident subscale of the Coping Styles Inventory.
Change in optimistic coping style | Baseline and 8 weeks after the intervention
  This secondary outcome measures changes in the use of optimistic coping strategies among caregivers after completing the Mindfulness-Based Self-Compassion Program. Measured by the optimistic subscale of the Coping Styles Inventory.
Change in seeking social support coping style | Baseline and 8 weeks post-intervention
  This outcome assesses whether participants demonstrate an increased tendency to seek social support as a coping strategy after participating in the program. Data will be collected via the social support subscale of the Coping Styles Inventory.
Change in helpless coping style | Baseline and 8 weeks after the intervention
  This outcome evaluates whether the program decreases the use of helpless coping strategies among participants. Assessed using the helpless subscale of the Coping Styles Inventory.
Change in submissive coping style | Baseline and 8 weeks after the intervention
  This outcome examines whether the intervention reduces submissive coping strategies among caregivers. It is measured by the submissive subscale of the Coping Styles Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Lök, Prof. Dr., Study Director — Selcuk University Faculty of Nursing
Locations (1):
- Selcuk University, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical concerns and privacy considerations. The study involves a sensitive population, and sharing such data is not deemed appropriate.